CLINICAL TRIAL: NCT03315533
Title: Altering The Transition From Acute to Chronic Pain (ATTAC-Pain): A Randomized Clinical Trial of Duloxetine for the Treatment and Prevention of Musculoskeletal Pain
Brief Title: Altering The Transition From Acute to Chronic Pain (ATTAC-Pain)
Acronym: ATTAC-PAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Mayday Fund (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RhodeIslandH
Record Dates: First submitted 2017-09-25; First posted 2017-10-20 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2018-12

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Duloxetine 30 milligrams (mg) (Experimental)
  Interventions: Drug: Duloxetine 30 milligrams (MG)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet
- Duloxetine 60 milligrams (mg) (Experimental)
  Interventions: Drug: Duloxetine 60 milligrams (MG)

INTERVENTIONS:
Drug: Duloxetine 30 milligrams (MG) — Once a patient's history and screening results have been cleared by a physician investigator, the participant will be randomized by the study site investigational drug services (IDS) to receive duloxetine (30mg or 60mg) vs. placebo
  Arms: Duloxetine 30 milligrams (mg)
Drug: Duloxetine 60 milligrams (MG) — Once a patient's history and screening results have been cleared by a physician investigator, the participant will be randomized by the study site investigational drug services (IDS) to receive duloxetine (30mg or 60mg) vs. placebo
  Arms: Duloxetine 60 milligrams (mg)
Drug: Placebo Oral Tablet — Once a patient's history and screening results have been cleared by a physician investigator, the participant will be randomized by the study site investigational drug services (IDS) to receive duloxetine (30mg or 60mg) vs. placebo
  Arms: Placebo

SUMMARY:
The current way that pain is treated after trauma and injury is problematic. Most often pain after trauma is treated with opioids (ex. Percocet® or Vicodin®) or anti-inflammatories (ex. ibuprofen). Both of these medications can cause side effects and opioids have been related to the development of addiction. In addition, there are not any treatments that prevent pain from going on to become persistent (last beyond it is supposed to) or chronic (lasting 3 months or longer).

Chronic pain is an enormous problem and there an urgent need to find both alternatives to opioid pain medications and medications that prevent pain from becoming chronic. The ATTAC-Pain (Altering The Transition from Acute to Chronic Pain) study proposes to examine whether duloxetine (a medication that is marketed for depression, anxiety, and specific types of pain conditions), can reduce acute and chronic pain among adults who come to the emergency department (ED)with muscular pain (such as neck pain after a car accident or low back pain). Investigators will enroll 60 patients who come to the ED. Patients will be eligible if they report moderate to severe muscular pain (such as pain in the back, neck, or shoulders). Consenting patients will be randomized to receive duloxetine 30mg, duloxetine 60mg, or placebo (2/3rd chance of being in one of the duloxetine groups). The study team will follow patients for six weeks and collect information on pain outcomes and use of pain medications. Investigators aim to determine if duloxetine can (1) reduce acute pain symptoms following the ED visit, (2) prevent the transition to persistent pain (having pain 6 weeks after the initial ED visit), and (3) decrease opioid use following a motor vehicle collision (MVC). The results of this study will ultimately help determine if duloxetine can be used as a non-opioid pain treatment option that reduces acute pain and prevents the transition to chronic pain. This in turn can improve recovery, reduce opioid use and its consequences, and decrease health care costs.

DETAILED DESCRIPTION:
There is an urgent need for new non-opioid pain management options to prevent the development of chronic musculoskeletal pain in patients experiencing acute pain and injury. Investigators propose to address this unmet need by intervening at the point when pain is still acute with pain management that is intended to alter the mechanisms involved in the transition from acute to chronic pain. The proposed study, "Altering The Transition from Acute to Chronic Pain (ATTAC-Pain): A randomized clinical trial of duloxetine for the treatment and prevention of musculoskeletal pain," will examine the ability of duloxetine to improve pain outcomes in individuals presenting to the emergency department (ED) with acute musculoskeletal pain. Investigators will enroll a total of sixty participants. Eligible patients who consent to the study will: be randomized in the ED, receive a dose of study drug (duloxetine 30mg, duloxetine 60mg, or placebo) in the ED, and be discharged from the ED with a two week supply of study drug. Following discharge, the patient will receive follow-up assessments via internet-based surveys and phone to monitor for adverse events and evaluate patient outcomes. The patient will also return to the study site for an in-person follow-up interview 6 weeks after their initial ED visit. The study team will recruit participants at the Rhode Island Hospital and the Miriam Hospital EDs. The results of this study will be used as basis for a potentially high impact large-scale trial examining an important new non-opioid pain treatment option that reduces acute pain and prevents the transition to chronic pain. This in turn can improve recovery, reduce opioid use and its sequelae, and decrease health care costs.

ELIGIBILITY:
Inclusion Criteria:

* generally in good health, are between the ages of 18 and 65, present to the ED with acute (present for <7 days) musculoskeletal pain, and have a current pain score of >4 without a history of pain in the past month.

Exclusion Criteria:

* Musculoskeletal pain lasting > 7days
* ED pain score <4
* Chronic pain: Pain present on most days of the week, with an average score >1 in past month, in the same location as presenting pain
* Clinically unstable
* Fracture (except fracture of the phalanges)
* Substantial soft tissue injury†
* Hepatic failure (acute or chronic)
* Renal failure (acute or chronic)
* Coronary artery disease, including previous myocardial infarction, Angina, percutaneous transluminal coronary angioplasty, etc.
* History of glaucoma
* Previous congestive heart failure
* History of seizure disorder
* History of mania or psychotic disorder
* History of suicidal ideation
* Prisoner
* History and behavior indicates, in the investigator's judgment, that the participant would likely be noncompliant with the study
* Any other condition that, in the investigator's judgment, would indicate that the patient in unsuitable for the study (e.g. might interfere with the study, confound interpretation, or endanger patient)
* Does not have a telephone
* Does not have regular internet access and email address
* Unable to speak and read English
* Blood pressure reading(s) in ED that, when considered in the context of patient past and current history, in the investigator's judgment exceeds acceptable level
* Currently taking a monoamine oxidase inhibitor (MAOI)
* Currently taking medication with substantial interaction with duloxetine (Table 1).
* Breastfeeding
* If female, either not postmenopausal (having menses within past year), or, if childbearing potential, positive pregnancy test prior to randomization and not using a medically acceptable form of contraception
* Exceeds acceptable chronic daily opioid use prior to MVC*
* Previously on duloxetine
* Previous allergic reaction to duloxetine
* Antidepressant use within 2 weeks of study start (4 week if Prozac)
* Allergy to lactose
* Intoxicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Self-reported axial pain (0 - 10 numeric rating scale) | through 6 weeks after enrollment visit
  Moderate to severe axial muscoloskeletal pain was chosen as the primary outcome because it is associated with risk for chronic pain development and because it of its clinical relevance. Investigators will asses if there is a decrease in persistent musculoskeletal pain incidence and severity 6 weeks after the ED visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beaudoin FL, Gaither R, DeLomba WC, McLean SA. Tolerability and efficacy of duloxetine for the prevention of persistent musculoskeletal pain after trauma and injury: a pilot three-group randomized controlled trial. Pain. 2023 Apr 1;164(4):855-863. doi: 10.1097/j.pain.0000000000002782. Epub 2022 Sep 15. PMID 36375173
- [Derived] Strauss DH, Santhanam DR, McLean SA, Beaudoin FL. Study protocol for a randomised, double-blind, placebo-controlled clinical trial of duloxetine for the treatment and prevention of musculoskeletal pain: altering the transition from acute to chronic pain (ATTAC pain). BMJ Open. 2019 Mar 5;9(3):e025002. doi: 10.1136/bmjopen-2018-025002. PMID 30842115